CLINICAL TRIAL: NCT01402934
Title: The Ability of Pulse Pressure Variation to Predict Fluid Responsiveness in Spontaneously Breathing Patients Undergoing Thoracic Surgery
Brief Title: Pulse Pressure Variation in Spontaneously Breathing Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Hyon Bahk, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JHBahk_PPV
Record Dates: First submitted 2011-05-29; First posted 2011-07-26 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2011-07

CONDITIONS: Pulse Pressure Variation; Spontaneously Breathing
MeSH Terms: interventions — HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- fluid infusion (Experimental)
  Interventions: Procedure: Hydroxyethyl starch solution (Voluven) infusion

INTERVENTIONS:
Procedure: Hydroxyethyl starch solution (Voluven) infusion — fluid loading will be performed by hydroxyethyl starch solution (Voluven), at 6 mL/kg

SUMMARY:
The investigators hypothesized that pulse pressure variation (PPV) could predict fluid responsiveness in spontaneously breathing patients undergoing anesthesia induction.

DETAILED DESCRIPTION:
Pulse pressure variation (PPV) is known to be a dynamic indicator to predict fluid responsiveness in mechanically ventilating patients. PPV is generated by cardiopulmonary interaction with respiratory cycles. In spontaneous breathing, the cardiopulmonary interaction may lead to PPV by inverted manner. In this study, the investigators will evaluate the ability of PPV to predict fluid responsiveness in spontaneously breathing patients. Before induction of anesthesia, radial artery cannulation is performed, and FloTrac/Vigileo (Edwards Lifesciences Corp., Irvine, USA) system is connected. And then, the investigators will measure baseline data including invasive blood pressure, pulse pressure, cardiac index, stroke volume variation in two different conditions: during tidal spontaneous breathing and during forced spontaneous breathing. All hemodynamic measurement will be repeated after infusion of fluid using 6mL/kg of hydroxyethyl starch solution (Voluven), and will be averaged over 3 minutes. Patients whose cardiac index increased by >15% to fluid infusion is defined as responders. The investigators will compare the hemodynamic parameters between responders and non-responders. To evaluate the ability to predict volume responsiveness, receiver operating characteristics curves of the PPV will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery

Exclusion Criteria:

* preoperative arrhythmia
* left ventricular ejection fraction <40%
* intra-cardiac valve disease
* intra-cardiac shunt
* pulmonary artery hypertension
* severe peripheral vascular obstructive disease
* decreased pulmonary function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
pulse pressure variation | three respiratory cycles, an expected average of 30 seconds

SECONDARY OUTCOMES:
hemodynamic parameters | before and after fluid loading, 1 mimute
  systolic blood pressure (SBP), dyastolic BP, mean BP, heart rate, cardiac index, stroke volume varation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea